CLINICAL TRIAL: NCT00605384
Title: A Comparative Study of the Antiviral Efficacy and Safety of Entecavir Plus Tenofovir Versus Adefovir Added to Continuing Lamivudine in Adults With Lamivudine- Resistant Chronic Hepatitis B Virus Infection
Brief Title: A Phase IIIb Study to Compare Entecavir Plus Tenofovir vs. Adefovir Added to Continuing Lamivudine Therapy in Adult Patients With Lamivudine-Resistant Hepatitis B Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Objectives Have Changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AI463-137
Record Dates: First submitted 2008-01-18; First posted 2008-01-31 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir; adefovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Entecavir + Tenofovir
- 2 (Experimental)
  Interventions: Drug: Adefovir + continuing Lamivudine

INTERVENTIONS:
Drug: Entecavir + Tenofovir — Tablets, Oral Entecavir 1 mg + Tenofovir 300 mg, once daily, 100 weeks
  Other Names: Baraclude
  Arms: 1
Drug: Adefovir + continuing Lamivudine — Tablets, Oral, Adefovir 10 mg + Lamivudine, 100 mg, once daily, 100 weeks
  Arms: 2

SUMMARY:
The purpose of this clinical research study is to find out whether a combination of entecavir (ETV) plus tenofovir (TNF) works better against Hepatitis B virus than adefovir (ADV) added to continuing lamivudine (LVD) therapy in patients whose Hepatitis B virus (HBV) is resistant against lamivudine. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HBV infection
* History of lamivudine (LVD) treatment, and lamivudine resistance (LVDr), receiving LVD at screening visit
* Compensated liver function
* HBV DNA ≥ 172,000 IU/mL
* Hepatitis B e-antigen (HBeAg)-positive or HBeAg-negative

Exclusion Criteria:

* Evidence of decompensated cirrhosis
* Coinfection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis D virus (HDV)
* Recent history of pancreatitis
* Serum alpha fetoprotein > 100 ng/mL
* Except lamivudine, any prior therapy with nucleoside or nucleotide analogue antiviral agents with activity against hepatitis B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (4):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - Rush University Medical Center, Chicago, Illinois
  - Local Institution, New York, New York
- Belgium (2):
  - Local Institution, Brussels
  - Local Institution, Leuven
- Germany (4):
  - Local Institution, Berlin
  - Local Institution, Bonn
  - Local Institution, Düsseldorf
  - Local Institution, Mainz
- Italy (5):
  - Local Institution, Messina
  - Local Institution, Modena
  - Local Institution, Naples
  - Local Institution, Padua
  - Local Institution, San Giovanni Rotondo
- Poland (3):
  - Local Institution, Chorzów
  - Local Institution, Krakow
  - Local Institution, Lublin
- Turkey (Türkiye) (6):
  - Local Institution, Ankara
  - Local Institution, Istanbul
  - Local Institution, Izmir
  - Local Institution, Kocaeli
  - Local Institution, Sihhiye Ankara
  - Local Institution, Trabzon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 84 subjects were to be treated with entecavir (ETV) plus tenofovir (TNF) or adefovir (ADV) added to continuing lamivudine (LVD).
Pre-assignment Details: Of the 4 subjects enrolled, 2 were not randomized (reasons: "Subject no longer meets study criteria" and "Other"). Both subjects randomized were treated as well.
Groups:
- Entecavir + Tenofovir: Tablets, Oral, Entecavir 1 mg + Tenofovir 300 mg, once daily, 100 weeks
Period: Overall Study
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Started | 1 | 1
Completed | 0 (study terminated early) | 0 (study terminated early)
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved an Hepatitis B Virus DNA (HBV DNA) Level < 50 IU/mL at Week 48
Description: using the Roche COBAS® TaqMan HBV Test for use with the High Pure System (HPS) assay, by Polymerase Chain Reaction (PCR); HBV DNA < 50 IU/mL = approximately 300 copies/mL
Time Frame: Week 48
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: Participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Who Achieved an HBV DNA Level <50 IU/mL at Week 96
Description: by PCR, using the Roche COBAS®TaqMan - HPS assay; HBV DNA < 50 IU/mL = approximately 300 copies/mL.
Time Frame: Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuations Due to AEs or Laboratory Abnormalities
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and/or is an important medical event.
Time Frame: Day 1 through end of treatment (Week 100 +/- 5 days)
Population: All treated participants. Timeframe for Outcome Measure revised due to study termination. (Study Completion Date=February 2009).
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 1 | 1
participants
  AEs | 1 | 1
  SAEs | 0 | 0
  Deaths | 0 | 0
  Discontinuations due to AEs | 0 | 0
  Discontinuations due to Laboratory Abnormalities | 0 | 0

4. Secondary Outcome: Number of Participants Who Achieved HBV DNA < the Lower Limit of Detection (LLD) at Weeks 48 and 96
Description: by PCR, using the Roche for the Roche COBAS® TaqMan - HPS assay. LLD = 4.8 IU/mL (approximately 28 copies/mL)
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: HBV DNA Values at Weeks 48 and 96
Description: Number of Participants with HBV DNA <LLD (4.8); LLD to <50; 50 to <172; 172 to <1,720; 1,720 to <17,200; and ≥17,200 IU/mL (<LLD (28); 28 to <300; 300 to <1,000; 1,000 to <10,000; 10,000 to <100,000; and ≥100,000 copies/mL by PCR, using the Roche COBAS®TaqMan - HPS assay
Time Frame: Weeks 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Mean log10 Reduction From Baseline in HBV DNA at Weeks 48 and 96
Description: by PCR, using the Roche COBAS®TaqMan - HPS assay
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints was analyzed.
Measure: Mean (Standard Deviation); unit: log10
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) > 1 x Upper Limit of Normal (ULN) at Baseline Who Achieved ALT Normalization (≤ 1 x ULN) at Weeks 48 and 96
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: Participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Who Were Hepatitis B E-antigen (HBeAg)-Positive at Baseline With Loss of HBeAg at Weeks 48 and 96
Description: HBeAg is a hepatitis B viral protein. It is an indicator of active viral replication.
Time Frame: Baseline, Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints was analyzed.
Measure: Number; unit: Participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Who Were HBeAg-positive at Baseline With HBe Seroconversion at Weeks 48 and 96
Description: HBe seroconversion = HBeAg loss and presence of hepatitis B e-antibody (HBeAb)
Time Frame: Baseline, Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Hepatitis-B-Virus Surface Antigen of the (HBsAg) Loss at Weeks 48 and 96
Description: Hepatitis B surface antigen (HBsAg) = a part of the hepatitis B virus that, when in the blood, is an early marker of infection
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Participants With HBs Seroconversion (HBsAg Loss and Presence of HBsAb) at Weeks 48 and 96
Description: Hepatitis B surface antigen (HBsAg) = a part of the hepatitis B virus that, when in the blood, is an early marker of infection. HBsAb = HBsAg antibodies. HBs Seroconversion = HBsAg loss and presence of HBseAb
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of Participants With Genotypic Resistance Based on Analysis of Samples From Participants With HBV DNA ≥ 50 IU/mL at Weeks 48 and 96
Description: HBV DNA ≥ 50 IU/mL = approximately 300 copies/mL
Time Frame: Week 48, Week 96
Population: Due to early study termination, none of the efficacy endpoints were analyzed.
Measure: Number; unit: participants
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Entecavir + Tenofovir | Adefovir + Continuing Lamivudine
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir + Tenofovir (N=1) | Adefovir + Continuing Lamivudine (N=1)
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Following review of business priorities, BMS decided to terminate this study at an early stage. This was a strategic decision, not based on clinical or safety concerns. Due to limited data, no conclusions on safety and efficacy can be made.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.